CLINICAL TRIAL: NCT06634836
Title: In-trial Qualitative Interviews to Explore the Impact of Gene Therapy in Hemophilia A & B
Brief Title: Patient Interview Study to Explore the Impact of Gene Therapy in Hemophilia A & B
Status: Withdrawn | Type: Observational
Why Stopped: Business decision
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3731011; NCT06634836 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-01; First posted 2024-10-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia A; Hemophilia B; Genetic Therapy
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemophilia A and Hemophilia B patients: Patients who are participating in the Pfizer's gene therapy clinical trials for Hemophilia A or Hemophilia B or are in the long-term follow up for these clinical programs

SUMMARY:
The purpose of this study is to learn about experiences of patients with hemophilia A and B after taking gene therapy. The experiences of patients will be studied through online interviews.

This study is seeking participants who are:

* part of the Pfizer's gene therapy clinical studies or
* in the long-term follow up for these clinical programs. Participants will have one study visit at the clinic and one online interview. The planned duration for each participant will be 1 to 2 months. This covers the time from entering the study to end of the online interview.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Pfizer's gene therapy clinical trials for Hemophilia A or B .
* Participants will be one year or more post-gene therapy
* Participants will be willing to provide written consent and will be willing to comply with the study requirements

Exclusion Criteria:

-No exclusion criteria

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who are participating in the Pfizer's gene therapy clinical trials for Hemophilia A and B or are in the long-term follow up for these clinical programs
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of self-reported symptoms pre and post hemophilia gene therapy | From date of dosing in the gene therapy clinical trial until the interview date, no less than 52 weeks.
Frequency of self-reported severity pre and post hemophilia gene therapy | From date of dosing in the gene therapy clinical trial until the interview date, no less than 52 weeks.
Frequency of self-reported impacts pre and post hemophilia gene therapy | From date of dosing in the gene therapy clinical trial until the interview date, no less than 52 weeks.
Change in the proportion of patients answering 5-point Likert scale questions about the burden of hemophilia on the participant's life pre-post gene therapy | From date of dosing in the gene therapy clinical trial until the interview date, no less than 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.